CLINICAL TRIAL: NCT01209052
Title: A Single-centre, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerabilty, Pharmacokinetics, and Pharmacodynamics of Single, Oral, Ascending Doses and Repeat Oral Doses of GSK1325756 in Healthy Male Subjects.
Brief Title: First Time in Human Study With GSK1325756
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 112483
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; CXCR2 inhibitor
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — danirixin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- COHORT 1 (Experimental): Interlocking design with Cohort 2. Single dose; treatment period over 2 days such that two subjects will receive GSK1325756 and at least one subject will receive placebo on Day 1. The remaining subjects will be dosed on day 2 of each treatment period assuming adequate safety from Day 1. Placebo and an escalation of GSK1325756 from 10mg, to 50mg, and 200mg, will be administered over the 6 week long treatment period allowing adequate washout period between doses.
  Interventions: Drug: GSK1325756; Other: Placebo
- COHORT 2 (Experimental): Interlocking design with Cohort 1. Single dose; treatment period over 2 days such that two subjects will receive GSK1325756 and at least one subject will receive placebo on Day 1. The remaining subjects will be dosed on day 2 of each treatment period assuming adequate safety from Day 1. Placebo and an escalation of GSK1325756 from 25mg, to 100mg, and 400mg, will be administered over the 6 week long treatment period allowing adequate washout period between doses.
  Interventions: Drug: GSK1325756; Other: Placebo
- COHORT 3 (Experimental): Placebo controlled, 14-day, once daily, repeat-dose evaluation with one selected dose of GSK1325756 in 14 subjects. Dose selection based on review of safety and tolerability data from cohorts 1 and 2.
  Interventions: Drug: GSK1325756; Other: Placebo
- COHORT 4 (Experimental): Placebo controlled, 14-day, once daily, repeat-dose evaluation with a higher selected dose of GSK1325756 in 14 subjects. Dose selection based on review of safety and tolerability data from cohort 3.
  Interventions: Drug: GSK1325756; Other: Placebo

INTERVENTIONS:
Drug: GSK1325756 — Drug will be orally administered in varying amounts over varying time periods as detailed in the 'arms' section.
Other: Placebo — Placebo will be orally administered to at least 4 subjects in each treatment period of each cohort. In each sequence in each cohort, all subjects will receive one dose of placebo.

SUMMARY:
This study aims to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of single, oral ascending doses, and repeat oral doses of GSK1325756 administered to healthy adult male volunteers. This study is the First Time in Human study for GSK1325756.

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability, pharmacokinetics(PK) and pharmacodynamics (PD) of single and repeat oral doses of GSK1325756 in healthy, male volunteer subjects, including the assessment of the effect of GSK1325756 on ex vivo 'C-X-C Motif Ligand 1' (CXCL1)-induced 'Cluster of Differentiation 11b' (CD11b) cell surface expression on peripheral blood neutrophils. Selective antagonism of the interaction between 'C-X-C Receptor Type 2' (CXCR2) and its various chemokine ligands provides a potential strategy for reducing the underlying inflammation that contributes to the progression of Chronic Obstructive Pulmonary Disease (COPD). This study is the first administration of GSK1325756 to humans and will be conducted in four cohorts.

Cohorts 1 and 2 will comprise of a double-blind, placebo-controlled, single dose escalation of GSK132576 in healthy adult males in two interlocking cohorts.

The data generated from this single dose escalation component of the study (safety, tolerability, and where applicable, PK profile, and, if available, PD data) will enable decisions regarding progression from one to dose the next higher dose later within Cohorts 1 and 2. This data will also be reviewed in decisions regarding study progression to repeat dosing in Cohorts 3 and 4, and the most suitable doses of GSK1325756 that should be selected for these repeat dose cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Aspartate Transaminase (AST), Alanine Transaminase (ALT), alkaline phosphatase and bilirubin ≤ 1.5x Upper Limit of Normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and Electrocardiogram (ECG). A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Males between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Subjects must agree to use one of the contraception methods listed below:

To prevent pregnancy in a female partner or to prevent exposure of any partner to the investigational product from a male subject's semen, male subjects must use one of the following contraceptive methods:

* Abstinence, defined as sexual inactivity consistent with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
* Condom (during non-vaginal intercourse with any partner - male or female) OR
* Condom and occlusive cap (diaphragm or cervical/vault caps) plus spermicidal agent (foam/gel/film/cream/suppository) (during sexual intercourse with a female) This criterion must be followed from the time of the first dose of study medication until at least 3-months post-last dose of study drug.

  * Body weight ≥ 60 kilograms (kg) and Body Mass Index (BMI) within the range 19 - 31 kilogrammes per square metre (kg/m-2) (inclusive)
  * 12-lead ECG without any clinically significant abnormality as judged by the Investigator, and average QTcB or QTcF (ECG paramaters) < 450 msec
  * Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
  * Able to complete all study procedures and planned treatment periods.

Exclusion Criteria:

* Cotinine or Exhaled Breath Carbon Monoxide (CO) Test indicative of current smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* A neutrophil count at screening of < 2 x 10(9) per litre (/L)
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Significant cardiac, pulmonary, metabolic, renal, gastrointestinal or other conditions that in the opinion of the investigator and/or GSK medical monitor, places the subject at an unacceptable risk as participant in this trial
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units for males. One unit is equivalent to 8 grams of alcohol: a half-pint (~240 milliLitres(mL)) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 3 months, 5 half-lives or twice the duration of the expected biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety. Prescription and non-prescription non-steroidal anti-inflammatory drugs are not permitted.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Subject is mentally or legally incapacitated.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-10-15 (Actual); Primary Completion 2010-03-02 (Actual); Study Completion 2010-03-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerabilty of GSK1325756 as assessed by clinical monitoring of blood pressure, pulse rate, ECG, and laboratory data, as well as reporting of AEs. | Study duration

SECONDARY OUTCOMES:
Area under the blood concentration-time curve, Maximum Concentration (Cmax), Time to Cmax (Tmax), terminal half-life and oral clearance of GSK1325756 following the administration of single escalating oral doses of GSK1325756 in healthy adult subjects. | Study duration
Area under the blood drug concentration-time curve, trough 24-hour Concentration (C24), Cmax, Tmax and accumulation of GSK1325756 following the administration of once daily repeat doses of two selected doses of GSK1325756 for 14 days in healthy subjects. | Study duration
Flow cytometric quantification of CXCL1-induced CD11b cell surface expression on peripheral blood neutrophils ex vivo following the administration of single and repeat oral doses of GSK1325756 in healthy adult subjects | Study duration
PK-PD model of the relationship between the blood concentration of GSK1325756 and CXCL1-induced CD11b cell surface expression on neutrophils ex vivo following the administration of single and repeat oral doses of GSK1325756 in healthy adult subjects | Study duration

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Miller BE, Mistry S, Smart K, Connolly P, Carpenter DC, Cooray H, Bloomer JC, Tal-Singer R, Lazaar AL. The pharmacokinetics and pharmacodynamics of danirixin (GSK1325756)--a selective CXCR2 antagonist --in healthy adult subjects. BMC Pharmacol Toxicol. 2015 Jun 20;16:18. doi: 10.1186/s40360-015-0017-x. PMID 26092545
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 112483 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/112483?search=study&search_terms=112483#rs
- Available data/document: Dataset Specification: 112483 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112483 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112483 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112483 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112483 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112483 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112483 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register